CLINICAL TRIAL: NCT04772807
Title: Validation of Kinocardiography, a New Technology Measuring Cardiac Mechanical Activity Via Accelerometers and Gyroscopes
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2020/502; Sponsor study reference (Other: FONDERASME_SRB2020340)
Record Dates: First submitted 2021-02-18; First posted 2021-02-26 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation; Hypertension; Heart Failure
MeSH Terms: conditions — Atrial Fibrillation; Hypertension; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- Healthy
  Interventions: Device: Kinocardiograph
- Patients infected by COVID- 19 with no symptoms
  Interventions: Device: Kinocardiograph
- Patients infected by COVID- 19 with symptoms
  Interventions: Device: Kinocardiograph
- Patients diagnosed with atrial fibrillation
  Interventions: Device: Kinocardiograph
- Hypertensive patients
  Interventions: Device: Kinocardiograph
- Heart failure patients, EF < 40%
  Interventions: Device: Kinocardiograph
- Heart failure patients, EF > 40% and < 60%
  Interventions: Device: Kinocardiograph
- Heart failure patients, EF > 60%
  Interventions: Device: Kinocardiograph

INTERVENTIONS:
Device: Kinocardiograph — Measure with the Kinocardiograph device and the Okcardio application installed on a smartphone
  Other Names: OKCARDIO smart application

SUMMARY:
Kinocardiographic measures mechanical and electrical function of the heart. The proposed solution is based on measurements of body vibrations. By measuring these movements on the surface of the body, it is possible to deduce, taking into account the individual's weight and size, the quality of the heartbeat that caused this vibration. The technique developed consists of a device measuring these vibrations at two places in the body: on the torso (Seismocardiography) and on the lower back (Ballistocardiography). The first measurement is a reflection of the local strength of the heartbeat as well as the transmission of blood to the body's main artery, the aorta. The second measurement, in the lower back, is the result of the contraction and movement of blood within the arterial system. Based on these two measurements, the energy produced by the heart and transmitted to the torso or the whole body is calculated. The energy over an entire cardiac cycle and the distribution of that energy within a heartbeat are used to characterize the mechanical function of the heart.

Clinical studies carried out previously have demonstrated the repeatability of kinocardiographic measurements (KCG) and their robustness with respect to the use of different sensors.

KCG measurements also showed a high sensitivity (> 94%) to different hemodynamic states induced by the injection of active inotropic agents, i.e. dobutamine also used as a treatment for heart failure in an advanced stage. In a randomized, double-blind, cross-over study controlled by Placebo, these measurements showed a strong correlation (r = 0.8, p <0.0001) with cardiac output measured by echocardiography. The technique has also demonstrated its ability to track changes in cardiac mechanical function during expiratory voluntary apnea.

KCG measurements were also evaluated during a micro-gravity simulation in Bedrest on 23 healthy volunteers. The measurements tracked cardiac deconditioning in the control group compared to the exercise group similarly to cardiac MRI measurements. Subsequently, KCG metrics showed an ability to distinguish reduced ejection fraction (HFrEF) heart failure patients from non-insufficient patients. These latest results also showed that the chest sensor alone was sufficient to separate HFrEF patients from normative patients, laying the foundation for possible use of the smartphone alone.

The prototype of a mobile application, named OKCARDIO, makes it possible to take measurements perfectly similar to the Kino thoracic sensor, but to date have never been used it in a clinical study. Such a tool would allow anyone with a smartphone-type mobile phone to measure their cardiac mechanical function themselves and make it available to the attending physician.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged above 18 years old.
* BMI (Body Mass Index) is below 50 kg/m2.
* Fit in one of the groups

Exclusion Criteria:

* Patients younger than 18 years old.
* BMI (Body Mass Index) higher than 50 kg/m2.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients in the ambulatory routine of the cardiology department at the Erasme hospital
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Feasibility of KCG measurement performed by the patients themselves | 12 weeks
  Feasibility is assessed by a repeatability score, namely the intraclass correlation coefficients ranging from 0, a non repeatable measure to 1 a perfectly repeatable measure .The score is computed between measure done at the hospital by a professional and the one done by the patient at the hospital and at home.
Validation of KCG parameters by comparisons from different modalities: Kinocardiograph device and OKCARDIO smartphone application. | Through study completion, an average of 1 year
Repeatability of OKCARDIO smartphone application recorded by an experimented operator and by the patient | Through study completion, an average of 1 year

SECONDARY OUTCOMES:
Compliance percentage of patients measuring KCG at home with the OKCARDIO smartphone application or the Kinocardiograph device. | 12 weeks
Mean and interquartile ranges of KCG derived HRV over the observation period. | Through study completion, an average of 1 year
  Mean and interquartile ranges of KCG derived HRV over the observation period in patients with active clinical syndromes that may be concomitant in the field of cardiac disorders (hypertension, atrial fibrillation, ischemia, valvulopathy, heart-failure,…) and pulmonary (asthma, infection,..). These clinical diagnoses are supported by the physical examination and the patient's medical record at inclusion.
Mean and interquartile ranges of KCG derived HR over the observation period. | Through study completion, an average of 1 year
  Mean and interquartile ranges of KCG derived HR over the observation period in patients with active clinical syndromes that may be concomitant in the field of cardiac disorders (hypertension, atrial fibrillation, ischemia, valvulopathy, heart-failure,…) and pulmonary (asthma, infection,..). These clinical diagnoses are supported by the physical examination and the patient's medical record at inclusion.
Adverse events related to the use of the Kinocardiograph devices and/or OKCARDIO smartphone. Count of adverse events. | Through study completion, an average of 1 year
Mean and interquartile ranges of KCG parameters (Kinetic Energy, namely iK) over the observation period. | Through study completion, an average of 1 year
Build a predictive score on a selection of several kinocardiography parameters based on machine learning algorithms with the aim to sort patients according to their pathological status. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Philippe van de Borne, Professor, Principal Investigator — Hospital Erasme
Locations (1):
- Erasme Hospital, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Hossein A, Mirica DC, Rabineau J, Rio JID, Morra S, Gorlier D, Nonclercq A, van de Borne P, Migeotte PF. Accurate Detection of Dobutamine-induced Haemodynamic Changes by Kino-Cardiography: A Randomised Double-Blind Placebo-Controlled Validation Study. Sci Rep. 2019 Jul 19;9(1):10479. doi: 10.1038/s41598-019-46823-3. PMID 31324831
- [Background] Rabineau J, Hossein A, Landreani F, Haut B, Mulder E, Luchitskaya E, Tank J, Caiani EG, van de Borne P, Migeotte PF. Cardiovascular adaptation to simulated microgravity and countermeasure efficacy assessed by ballistocardiography and seismocardiography. Sci Rep. 2020 Oct 19;10(1):17694. doi: 10.1038/s41598-020-74150-5. PMID 33077727
- [Background] Hossein A, Rabineau J, Gorlier D, Del Rio JIJ, van de Borne P, Migeotte PF, Nonclercq A. Kinocardiography Derived from Ballistocardiography and Seismocardiography Shows High Repeatability in Healthy Subjects. Sensors (Basel). 2021 Jan 26;21(3):815. doi: 10.3390/s21030815. PMID 33530417
- [Background] Morra S, Hossein A, Rabineau J, Gorlier D, Racape J, Migeotte PF, van de Borne P. Assessment of left ventricular twist by 3D ballistocardiography and seismocardiography compared with 2D STI echocardiography in a context of enhanced inotropism in healthy subjects. Sci Rep. 2021 Jan 12;11(1):683. doi: 10.1038/s41598-020-79933-4. PMID 33436841